CLINICAL TRIAL: NCT04245267
Title: Effect of Multicomponent Integrated Care Intervention on the Metabolic Control and Quality of Life in Patients With Type 2 Diabetes: the Mexico City DIAbetes EMPowerment and Improvement of Care Program
Brief Title: Multicomponent Integrated Intervention on Metabolic Control and Quality of Life in Type 2 Diabetes: DIABEMPIC Program
Acronym: DIABEMPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Especializada en el Manejo de la Diabetes en la Ciudad de Mexico (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIABEMPIC Mexico City
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes outcomes; glycemic control; self-care; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The effect of the intervention will be determined on the improvement on metabolic parameters, as well as in self care activities and quality of life using a "before and after" design. As a secondary analysis, results will be compared with the population in the wait-list receiving routine care in primary care units. Subjects who attend Clinica Especializada en el Manejo de la Diabetes and meet the selection criteria will be included in this study. Once their admission to the study is decided, subjects may participate in the recruitment and intervention stage and then in the annual follow-up visit stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the wait-list being attended with the standard model of care for diabetes in primary care units.
- DIABEMPIC program (Experimental): Intervention comprised by an interdisciplinary team care, patient-centered care approach, structured diabetes education program, promotion of self-management, audit, and guaranteed supply of anti-diabetic medication.
  Interventions: Behavioral: DIABEMPIC

INTERVENTIONS:
Behavioral: DIABEMPIC — Patients are attended by 9 diabetes health-care professionals every 2 weeks for 5 months in a shared medical appointment scheme, including individual and group sessions. Patients will be evaluated at the end of the program and 1 year after.
  Arms: DIABEMPIC program

SUMMARY:
Type 2 diabetes is one of the leading causes of morbidity and mortality rate in Mexico. Although important advances in treatment strategies have been developed in type 2 diabetes mellitus, large gaps exist in achieving quality of care. Few studies have determined the effect of multicomponent interventions in low and middle income countries. The DIABEMPIC program is a quality of care initiative developed by primary care public health services of the Mexico City Government to propitiate diabetes empowerment in people living with type 2 diabetes through an intervention comprised by an interdisciplinary team care, shared medical appointment scheme, patient-centered care approach, structured diabetes education program, promotion of self-management, audit, and guaranteed supply of anti-diabetic medication. The DIABEMPIC program target population consists of patients with type 2 diabetes, without advanced chronic complications, who have regular care in the public primary care services in Mexico city.

DETAILED DESCRIPTION:
Background: Diabetes mellitus is a chronic metabolic disease with disabling, deadly, and costly consequences for individuals, families, and national health care systems. Proper diabetes management in people living with type 2 diabetes mellitus focuses on reducing the risks for macrovascular and microvascular complications through controlling blood pressure, lipid levels, and blood glucose levels, and avoiding tobacco. Although important advances in pharmacological and non-pharmacological strategies have been developed, large gaps exist in achieving care goals, particularly in real-world practice and low- and middle- income countries. Barriers to care in T2DM patients may include lack of medical care, poverty, long distances or lack of time to get medical attention, lack of confidence, and inadequate social support, among others. Achievement of diabetes care goals: normal glycated hemoglobin, blood pressure, and LDL cholesterol is associated with better health outcomes, including lower risks of complicating events and death. The DIABEMPIC program is a quality of care initiative developed by primary care public health services of the Mexico City Government to propitiate diabetes empowerment in people living with type 2 diabetes through a 6-months intervention comprised by an interdisciplinary team care, shared medical appointment scheme, patient-centered care approach, structured diabetes education program, promotion of self-management, audit, , and guaranteed supply of anti-diabetic medication. The DIABEMPIC program target population consists of patients with type 2 diabetes, without advanced chronic complications, who have regular care in the public primary care services in Mexico city.

Hypothesis: Participation in the Diabetes Empowerment and Improvement of Care strategy allows reaching diabetes care goals.

General objective: To quantify diabetes care goals achievement at the end of the intervention and one year after finishing the comprehensive care program designed to propitiate diabetes empowerment at Clínica Especializada en el Manejo de la Diabetes of the Mexico City Government.

Specific objectives: To measure the program impact through the following variables: glycated hemoglobin, blood lipids, arterial pressure, self-care activities, diabetes knowledge, health related quality of life, incidence of complications and use of hospital services.

Goals: To improve diabetes care through this multicomponent intervention in order to prevent complications and and enhance quality of life in people with diabetes, but also to expand the care model to primary care health units in Mexico City.

Methodology: The DIABEMPIC program is a quality of care initiative developed by primary care public health services of the Mexico City Government to propitiate diabetes empowerment in people living with type 2 diabetes through an intervention comprised by an interdisciplinary team care, shared medical appointment scheme, patient-centered care approach, structured diabetes education program, promotion of self-management, audit, and guaranteed supply of anti-diabetic medication. Intervention consists of visits at Clínica Especializada en el Manejo de la Diabetes to attend individual and group sessions in a shared medical appointment model by an interdisciplinary case management team. The program last five months and visits occur every 2 weeks according to the needs assessed by the interdisciplinary team. Interdisciplinary team include: endocrinology, diabetes educator, nutritionist, podiatrist, ophthalmologist, psychologist, social worker and dentist. At each visit standardized interventions based in clinical practice guidelines are executed. At the initial, last visit and yearly visit preset indicators are evaluated, including: weight, blood pressure, glycated hemoglobin, lipid profile, creatinine, albumin/creatinin index in urine sample and validated questionaires related to diabetes self-care (Summary of Diabetes Self-care Activities) and Health related quality of life (EuroQOL-5Q-5L). The effect of the intervention will be determined on the improvement on metabolic parameters, as well as in self care activities and quality of life using a "before and after design". As a secondary analysis, results will be compared with the population in the wait-list receiving routine care in primary care units.

Expected results: In case of demonstrating its effectiveness, DIABEMPIC program is considered to be expanded in order to allow more people living with diabetes to receive the benefits of a Multicomponent intervention in Mexico City.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Older than 18 years old, younger than 70 years old
* Having diagnosis of type 2 diabetes
* Acceptance for participation in the program by signing informed consent sheet

Exclusion Criteria:

* Any other type of diabetes, such as Type 1 diabetes, LADA type Diabetes, gestational diabetes, or any other type of diabetes related to genetic syndromes
* advanced diabetes complications such as ischemic heart disease, NYHA III-IV heart failure, KDOQI renal failure ≥4, cerebral vascular disease with functional sequelae
* those who have comorbidities that limit their life expectancy such as malignant tumors in advanced stages
* Dependence of illicit drugs
* Conditions that require short-term surgical treatment.
* Advanced cognitive deficit or serious psychiatric disorders that hinder treatment adherence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-01-07 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control after the program | 5 months
  HbA1c (%): HbA1c will be compared from the first visit with the last visit (5 months later)

SECONDARY OUTCOMES:
Glycemic control after 1 year | 1 year
  HbA1c (%): HbA1c will be compared from the the last visit with the visit 1 year apart
Lipid control | 5 months
  Total Cholesterol, HDL-Cholesterol and Non-HDL Cholesterol in mg/dL will be compared from the first visit with the last visit (5 months later).
Weight change | 5 months
  Weight Change (Kg) will be compared from the first visit with the last visit (5 months later).
Blood pressure | 5 months
  Systolic and diastolic blood pressure (mmHg) will be compared from the first visit with the last visit (5 months later).
Blood pressure | 1 year
  Systolic and diastolic blood pressure (mmHg) will be compared from the last visit with the visit 1 year apart.
Lipid control | 1 year
  Total Cholesterol, HDL-Cholesterol and Non-HDL Cholesterol in mg/dL will be compared from the last visit with the visit 1 year apart.
Weight change | 1 year
  Weight Change in kilograms will be compared from the last visit with the visit 1 year apart.
Summary of Self-care Activities (0-7, higher score means better self-care) | 5 months
  Summary of Self-care Activities Questionnaire (nutrition, exercise, glucose test, foot care) in days a week (0-7, higuer score means better self-care). Self-care will be compared from the first visit with the last visit (5 months later).
Summary of Self-care Activities (0-7, higher score means better self-care) | 1 year
  Summary of Self-care Activities Questionnaire (nutrition, exercise, glucose test, foot care) in days a week (0-7, higuer score means better self-care). Self-care will be compared from the last visit with the visit one year apart
Health-related Quality of Life perception assessed by EQ-5D Visual Analogue Scale questionnaire (0-100, higuer score means better Quality of life perception) | 5 months
  Health-related Quality of life perception with EQ-5D questionnaire visual analogue scale (0-100, higher score means better self-care). Health-related Quality of Life will be compared from the first visit with the last visit (5 months later).
Health-related Quality of Life perception assessed by EQ-5D Visual Analogue Scale questionnaire (0-100, higher score means better Quality of life perception) | 1 year
  Health-related Quality of life perception with EQ-5D questionnaire visual analogue scale (0-100, higuer score means better quality of life). Health-related Quality of Life will be compared from the last visit with the visit one year apart.
Health-related Quality of Life perception assessed by EQ-5D Indexed score (0-1, higher score means better Quality of life perception) | 5 months
  Health-related Quality of life perception with EQ-5D questionnaire indexed score (0-100, higuer score means better quality of life). Health-related Quality of Life will be compared from the first visit with the last visit (5 months later)
Health-related Quality of Life perception assessed by EQ-5D Indexed score (0-1, higher score means better Quality of life perception) | 1 year
  Health-related Quality of life perception with EQ-5D questionnaire indexed score (0-100, higuer score means better quality of life). Health-related Quality of Life will be compared from the last visit with visit one year apart

OTHER OUTCOMES:
Glycemic control of the patients who attended the program compared with patients attended in primary care units (wait-list) | 5 months
  HbA1c (%). Comparison will be the mean deviation change of patients attending the program and patients with routine care in 5 months follow-up.
Lipid control of the patients who attended the program compared with patients attended in primary care units (wait-list) | 5 months
  Total Cholesterol, HDL-Cholesterol and Non-HDL Cholesterol in mg/dL . Comparison will be the mean deviation change of patients attending the program and patients with routine care in 5 months follow-up.
Weight change of the patients who attended the program compared with patients attended in primary care units (wait-list) | 5 months
  Weight change in kilograms. Comparison will be the mean deviation change of patients attending the program and patients with routine care in 5 months follow-up.
Blood pressure of the patients who attended the program compared with patients attended in primary care units (wait-list) | 5 months
  Systolic and diastolic blood pressure change in mmHg. Comparison will be the mean deviation changes of patients attending the program and patients with routine care in 5 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Silva-Tinoco, Principal Investigator — Clínica Especializada en Manejo de la Diabetes Gobierno de Ciudad de México
Locations (1):
- Clínica Especializada en el Manejo de la Diabetes de la Ciudad de México from the Ministry of Health of the Mexico City Government, Mexico City, Iztapalapa, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data generated is not publicly available due that data used are from patients and are under policies for private confidential information, but will be available at the end of the study on reasonable request and using unidentifiable IDs. Results are planned to be shared through Journal publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2021. Available for 3 years.
Access Criteria: Undefined

REFERENCES:
- [Background] Aschner P, Gagliardino JJ, Ilkova H, Lavalle F, Ramachandran A, Mbanya JC, Shestakova M, Chantelot JM, Chan JCN. Persistent poor glycaemic control in individuals with type 2 diabetes in developing countries: 12 years of real-world evidence of the International Diabetes Management Practices Study (IDMPS). Diabetologia. 2020 Apr;63(4):711-721. doi: 10.1007/s00125-019-05078-3. Epub 2020 Jan 4. PMID 31901950
- [Background] Lim LL, Lau ESH, Kong APS, Davies MJ, Levitt NS, Eliasson B, Aguilar-Salinas CA, Ning G, Seino Y, So WY, McGill M, Ogle GD, Orchard TJ, Clarke P, Holman RR, Gregg EW, Gagliardino JJ, Chan JCN. Aspects of Multicomponent Integrated Care Promote Sustained Improvement in Surrogate Clinical Outcomes: A Systematic Review and Meta-analysis. Diabetes Care. 2018 Jun;41(6):1312-1320. doi: 10.2337/dc17-2010. PMID 29784698
- [Background] Basto-Abreu A, Barrientos-Gutierrez T, Rojas-Martinez R, Aguilar-Salinas CA, Lopez-Olmedo N, De la Cruz-Gongora V, Rivera-Dommarco J, Shamah-Levy T, Romero-Martinez M, Barquera S, Lopez-Ridaura R, Hernandez-Avila M, Villalpando S. [Prevalence of diabetes and poor glycemic control in Mexico: results from Ensanut 2016.]. Salud Publica Mex. 2020 Jan-Feb;62(1):50-59. doi: 10.21149/10752. Spanish. PMID 31869561